CLINICAL TRIAL: NCT00275353
Title: Effectiveness of an Individualized Symptom Education Program (ISEP) on the Symptom Distress of Women Receiving Radiation for Gynecological Cancer.
Brief Title: Effectiveness of an Individualized Symptom Education Program (ISEP)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: Canadian Cancer Trials Group (Network)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 9848; 014144; 14927; 12048; 266-2003; 03-0487-CE
Record Dates: First submitted 2006-01-10; First posted 2006-01-11 (Estimated); Last update posted 2006-05-26 (Estimated); Status verified 2006-01

CONDITIONS: Uterine Cancer; Cervical Cancer; Vaginal Cancer; Vulvar Cancer
MeSH Terms: conditions — Uterine Neoplasms; Uterine Cervical Neoplasms; Vaginal Neoplasms; Vulvar Neoplasms

INTERVENTIONS:
Behavioral: Individualized Symptom Education

SUMMARY:
The purpose of this study is to examine whether an Individualized Symptom Education Program (ISEP) is helpful to women to manage their symptoms when they are receiving radiation therapy for gynecological cancer.

It is expected that women who participate in the ISEP program will be better able to manage their symptoms and exprience less distress than women who receive usual care.

DETAILED DESCRIPTION:
Women who have radiation therapy for gynecological cancer may experience a number of symptoms including fatigue, pain, nausea, pelvic symptoms (urgent and frequent urination and bowel movements, vaginal discharge, vaginal itching, skin irritation), anxiety and depression. We know that individualized education programs have helped people with other types of cancer to better manage their symptoms, and we would like to find out whether such interventions are helpful to women with gynecological cancers.

This study will compare two types of education: 1) the symptom education program currently in place (usual care), and 2) an individualized symptom education program (ISEP). This study is being conducted because we do not know if one type of education in patients who receive radiation for gynecological cancers is better than the other. Both types of education are are described below.

Usual care: Usual symptom education during radiation treatment consists of receiving verbal and written education from a radiation oncologist, nurse and radiation therapist, and other members of the interdisciplinary team. The radiation therapist will see the patient everyday during her radiation treatment and her doctor and nurse will see her on a weekly basis. The patient will also see other members of the team, such as a dietitian and social worker as required.

Individualized symptom education: Individualized symptom education will include usual symptom education and also an education program that focuses on symptom management. The patient will meet with an advanced practice nurse on a weekly basis for six sessions of about 30 minutes each. The advanced practice nurse will ask about the symptoms the paient is experiencing and those that are most bothersome to her. She will be given information about specific strategies to manage those symptoms, including written education materials. These strategies will be based on published best practice guidelines.

Data on symptom experience will be collected at 3 points: at baseline, after completion of the education program (end of external beam treatment), and at 3 months following completion of the education program (3 months following completion of external radiation treatment).

ELIGIBILITY:
Inclusion Criteria:

* First time diagnosis of cancer of the uterus, cervix, vagina, or vulva
* Beginning first time radical radiation therapy to the pelvis of at least 4000cGy (with or without brachytherapy after external beam treatment and with or without concurrent chemotherapy)
* At least 18 years of age and over
* Able to speak and understand English

Exclusion Criteria:

* Receiving palliative cancer treatment
* Receiving split course radiation treatment
* Ovarian cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144
Dates: Start 2003-07; Study Completion 2006-02

PRIMARY OUTCOMES:
Symptom distress - measured by the Symptom Distress Scale (SDS) at baseline, end of treatment, and three (3) months post treatment.

SECONDARY OUTCOMES:
All secondary outcomes measured at baseline, end of treatment, and three (3) months post treatment.
Pain - measured by the Brief Pain Inventory-Short Form (BPI-SF)
Fatigue - measured by the Brief Fatigue Inventory (BFI).
Nausea - measured by the nausea subscale (items 4, 5, 7) on the Rhodes Index of Nausea and Vomiting (INVR)
Mood symptoms - measured by the Hospital Anxiety and Depression Scale (HADS).
Pelvic symptoms - measured by the Pelvic Symptom Index (PSI)

CONTACTS AND LOCATIONS:
Overall Officials: Karima Velji, RN, MSc, AOCN, PhD(C), Principal Investigator — University of Toronto
Locations (1):
- Princess Margaret Hospital; Toronto Sunnybrook Reginal Cancer Centre, Toronto, Ontario, Canada